CLINICAL TRIAL: NCT00985231
Title: Performance Evaluation of Contact Lenses Among a Population of Adapted Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 630
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Results first posted 2011-03-14 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Vision Disorders
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PureVision Multi-Focal contact lenses (Experimental)
  Interventions: Device: PureVision Multi-Focal contact lenses
- SofLens59 contact lens (Active Comparator)
  Interventions: Device: SofLens59 contact lens

INTERVENTIONS:
Device: PureVision Multi-Focal contact lenses — Contact lenses to be worn on a daily wear basis for 2 weeks.
  Arms: PureVision Multi-Focal contact lenses
Device: SofLens59 contact lens — Contact lenses to be worn on a daily wear basis for 2 weeks.
  Arms: SofLens59 contact lens

SUMMARY:
This study is being conducted to evaluate Bausch & Lomb PureVision Multi-Focal contact lenses compared to the Bausch & Lomb SofLens59 contact lens when worn by adapted soft contact lens wearers on a daily wear basis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have clear central corneas and be free of any anterior segment disorders.
* Subjects must be adapted soft contact lens wearers and agree to wear the study lenses on a daily wear basis for at least eight hours a day for approximately two weeks.
* Subjects must wear a lens in each eye and each lens must be of the same manufacture and brand.

Exclusion Criteria:

* Subjects participating in any drug or device clinical investigation within two weeks prior to entry into this study and/or during the period of study participation.
* Subjects with any systemic disease affecting ocular health
* Subjects with an active ocular disease or using any ocular medication.
* Subjects who have had any corneal surgery (eg, refractive surgery).

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 272 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly J Barna, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 25 sites, by 25 Investigators in the United States (US). First participant enrollment was 09/28/2009 and last participant exited the study 11/09/2009
Pre-assignment Details: 272 participants (544 eyes) were enrolled in the study, 7 participants were ineligible at baseline, 265 participants were eligible. 259 participants (518 eyes) completed the study.
Period: Overall Study
Arm/Group | PureVision Multi-Focal Contact Lenses | SofLens59 Contact Lens
Started | 133 | 132
Completed | 130 | 129
Not Completed | 3 | 3
Not completed — ineligible | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Study related symptoms & complaints | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PureVision Multi-Focal Contact Lenses | SofLens59 Contact Lens | Total
Number analyzed (Participants) | 133 | 132 | 265
Age, Customized [Number; unit: participants]
  30-35 years of age | 68 | 67 | 135
  36 -40 years of age | 65 | 65 | 130
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 97 | 211
  Male | 19 | 35 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 7 | 11 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 14 | 29
  White | 110 | 104 | 214
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Distance Visual Acuity (VA) Between Test and Control Lenses Worse Than 20/40.
Description: Eyes with distance lens VA of 20/40 or worse at study exit between test and control lenses.
Time Frame: 2 weeks
Population: All Eligible, Dispensed Eyes with non-missing scores
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PureVision Multi-Focal Contact Lenses | SofLens59 Contact Lens
Number analyzed (Participants) | 130 | 132
Number analyzed (eyes) | 260 | 257
eyes | 2 | 0

2. Secondary Outcome: Subjective Ratings of Eye Strain
Description: Convergence Insufficiency Symptom Survey (CISS), was used to assess eye strain symptoms measured on a scale of 1-4. 0 score=never, 4 score=always
Time Frame: 2 week visit
Population: All Eligible, Dispensed Eyes, CISS Composite Score
Measure: Mean (Standard Deviation); unit: CISS Composite Score
Arm/Group | PureVision Multi-Focal Contact Lenses | SofLens59 Contact Lens
Number analyzed (Participants) | 133 | 131
CISS Composite Score | 9.9 (9.6) | 9.0 (9.5)

ADVERSE EVENTS:
Time Frame: At each visit for 2 weeks
Description: There were no adverse events reported during the study. There were no events requiring medical treatment related to the Test lens
Arm/Group | PureVision Multi-Focal Contact Lenses | SofLens59 Contact Lens
Serious Adverse Events (participants affected / at risk) | 0/270 | 0/274
Other Adverse Events (participants affected / at risk) | 0/270 | 0/274

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study data generated as a result of this study will be regarded as confidential, until appropriate analysis and review by the Sponsor or its designee and the Investigator(s) are completed. The results of the study may be published or presented by the Investigator(s)after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.